CLINICAL TRIAL: NCT05318625
Title: A Prospective Study to Evaluate the Clinical Performance and Safety of the SIRIUS Endoscope System in Laparoscopic Gynecological Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Precision Robotics (Hong Kong) Limited (Industry)
Collaborators: Gleneagles Hospital (Other); Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRHK02_TD8072
Record Dates: First submitted 2022-03-25; First posted 2022-04-08 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Ovarian Cancer; Cervical Cancer; Gynecologic Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gynaecological laparoscopic surgery (Experimental): Eligible women aged 18 - 70 years, regardless of parity, who need laparoscopic gynaecological surgery and who provide informed consent prior to surgery
  Interventions: Device: Gynaecological laparoscopic surgery (Sirius System)

INTERVENTIONS:
Device: Gynaecological laparoscopic surgery (Sirius System) — The laparoscopic procedures were done in the usual manner. The only difference was for the study participants, the Sirius System was used in place of the usual conventional laparoscope. All other procedures and instruments including the number of ports remained the same.
  For every procedure using the Sirius System, a conventional laparoscope was on immediate standby to replace the Sirius System should there be an unanticipated equipment failure so that the procedure could be completed without delay.

SUMMARY:
Precision Robotics' Sirius Robotic Flexible Endoscopic System is a new fully integrated compact 3D laparoscopic camera system with a disposable single-use flexible tip that can change its viewing direction.

A Prospective Study to Evaluate the Clinical Performance and Safety of the SIRIUS Endoscope System in Laparoscopic Gynecological Surgery.

The study is a single-arm prospective study to evaluate the Performance and Safety of the SIRIUS Endoscope System.

DETAILED DESCRIPTION:
Minimally invasive surgery (MIS) is well established in gynecological surgery. Compared to laparotomy, MIS is associated with reduced morbidity and quicker recovery. With advancement in laparoscopic technology and techniques, MIS in gynecology has progressed from multi-port to single incision laparoscopic surgery (SILS) and vaginal natural orifice transluminal endoscopic surgery (vNOTEs), thus further reducing morbidity and enhancing recovery.

One of the challenges of MIS is the restriction of the range of surgical movement. To overcome these technical challenges, articulated instruments are increasingly being used. The SIRIUS Endoscope System is a new, fully integrated compact 3D laparoscopic camera system with a disposable single-use flexible tip that can change its viewing direction. The articulated tip has three degrees of freedom, enabling C and S-shaped bending, and providing a wider field of view compared to conventional laparoscopes. This wider field of view is of advantage for SILS and vNOTEs. Presently available commercial systems do not have the same field of view or degrees of freedom.

A first in-human, proof of concept, and early development study of the SIRIUS Endoscope System was done at GHK in 2021 (HKU-GHK IRB 2021-01, ClinicalTrials.gov NCT05048407). The successful completion of 11 of 13 (85%) planned procedures in this sequentially reported, prospective case series, shows that the SIRIUS Endoscope System can be used with indications of safety, and efficacy for intermediate and major MIS laparoscopic procedures in gynecology. The findings have been submitted for consideration for publication.

Based on the outcome of this study, further improvements to the SIRIUS Endoscope System have been made to enhance safety, reliability, and usability. This proposed prospective study is a confirmatory study to evaluate the performance and safety of the SIRIUS Endoscope System in preparation for regulatory approval.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are planned for Laparoscopic Gynecological Surgery (LGS)
* Patient is 18 years of age or older
* Signed written informed consent.

Exclusion Criteria:

* Patient is pregnant, or planning on becoming pregnant
* Obese patients (BMI >35)
* Patient with known contraindication(s) to Laparoscopic Gynecological Surgery
* Patient with operations planned for longer than 4 hours
* Subjects are considered ineligible for the study as judged by the investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women-only
Enrollment: 30 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
General Assessment of SIRIUS Endoscope System. | Through study completion, Up to 1 year from the first to the last patients
  General Assessment of SIRIUS Endoscope System, using Questionnaire- Clinical Study General Assessment of SIRIUS Endoscope System)
SIRIUS Endoscope Articulated tip assessment. | Through study completion, Up to 1 year from the first to the last patients
  SIRIUS Endoscope Articulated tip assessment, using the Questionnaire -Clinical Study Assessment of SIRIUS Endoscope System Articulated Tip

SECONDARY OUTCOMES:
The time of straight and bending positions of SIRIUS Endoscope System articulated tip | Through study completion, Up to 1 year from the first to the last patients
Events of device deficiency and/or malfunctions of SIRIUS Endoscope System | Through study completion, Up to 1 year from the first to the last patients
Intraoperative adverse events related to the SIRIUS Endoscope System | Through study completion, Up to 1 year from the first to the last patients
Postoperative complications related to the SIRIUS Endoscope System | Through study completion, Up to 1 year from the first to the last patients

CONTACTS AND LOCATIONS:
Overall Officials: Tong Yow Ng, MD, Principal Investigator — Gleneagles Hospital
Locations (1):
- Gleneagles Hospital Hong Kong, Wong Chuk Hang, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: First in-human trial and prospective case series of an articulated laparoscopic camera system in minimally invasive surgery in gynecology: an IDEAL stage 1 and 2a study — https://sit.bmj.com/content/bmjsit/4/1/e000117.full.pdf